CLINICAL TRIAL: NCT00088062
Title: A Phase I/IIa Trial of STA-5326 in Crohn's Disease Patients With CDAI Scores of 220-450
Brief Title: STA-5326 in Crohn's Disease Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5326-03; Crohn's Disease; CDAI Scores of 220-450
Record Dates: First submitted 2004-07-19; First posted 2004-07-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — apilimod

INTERVENTIONS:
Drug: STA-5326

SUMMARY:
The purpose of this study is to determine the safety and tolerability of STA-5326 given once daily or twice daily to Crohn's Disease patients with moderate disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years old
* Crohn's Disease for 6 months
* CDAI scores between 220-450
* +/- 5-ASA, stable dose for > 2 weeks
* +/- Corticosteroids, less than or equal to 40 mg per day with a stable dose for 2 weeks
* +/- Infliximab with no treatment within 4 weeks
* +/- 6-Mercaptopurine, with a stable dose for 8 weeks
* +/- Antibiotics, with a stable dose for 2 weeks

Exclusion Criteria:

* Patients who have had methotrexate, cyclosporine, or other experimental drug within 3 months of screening
* Pregnancy, breast feeding
* History of total proctocolectomy with stoma. Previous ileocolectomy would not be a contraindication to the study
* Bowel obstruction
* Surgical bowel resection within 90 days
* Total parenteral nutrition (TPN), CYA, tacrolimus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-02; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Venture Research Institute, LLC, North Miami Beach, Florida
  - Shafran Gastoenterology Center, Winter Park, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Heart of America Research Institute, Topeka, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Long Island Clinical Research, Great Neck, New York
  - Rochester Institute for Digestive Diseases and Sciences, Inc, Rochester, New York
  - Carolina Research Associates, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - West Hills GI, Portland, Oregon
  - Blair Gastroenterology Associates, Altoona, Pennsylvania
  - Memphis Gastroenterology Group, Memphis, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee